CLINICAL TRIAL: NCT07263048
Title: PrEP & Soccer: A Program for Pharmacy Chains to Increase PrEP Awareness and Access Among Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Mariano Juan Kanamori Nishimura, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20250645; 1R01AI191576-01 (NIH)
Record Dates: First submitted 2025-12-02; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: HIV Prevention; Latino Men Who Have Sex With Men; Pharmacy

STUDY DESIGN:
Intervention Model Description: 8 pharmacies randomized 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP & Soccer Intervention (Experimental): Pharmacies assigned to "PrEP & Soccer" group will receive personalized PrEP navigation support from the PrEP Navigator.
  Interventions: Behavioral: PrEP & Soccer PrEP Navigation
- Standard of care (CVS standard health information) (Active Comparator): Pharmacies assigned to the control group will receive a brochure describing services offered by CVS Health and the MinuteClinic.
  Interventions: Behavioral: CVS Health brochure

INTERVENTIONS:
Behavioral: PrEP & Soccer PrEP Navigation — Pharmacies assigned to this group will receive personalized PrEP navigation support provided by a PrEP Navigator following baseline assessment. Sessions may be brief (~15 minutes) or longer depending on participant needs. The navigator supplies a pamphlet describing PrEP (how it works, payment options), and CVS-provided HIV services; discusses whether PrEP or another HIV prevention strategy is best for the participant; and, if PrEP is selected, provides a referral to a PrEP provider.
  Arms: PrEP & Soccer Intervention
Behavioral: CVS Health brochure — Standard health information delivered via brochure, no active navigation components. Content includes a brochure describing services offered by CVS Health and the MinuteClinic.
  Arms: Standard of care (CVS standard health information)

SUMMARY:
This type 3 Hybrid Effectiveness-Implementation study will evaluate PrEP & Soccer, a multicomponent and multilevel implementation strategy delivered by a pharmacy chain to increase PrEP knowledge and initial PrEP appointment attendance among men. Using mixed methods and implementation science approaches, this parallel cluster randomized controlled study will assess key implementation factors at CVS Health pharmacy locations assigned either to the PrEP & Soccer intervention or to a general CVS Health service information-only control.

ELIGIBILITY:
Inclusion Criteria:

* Provide their informed consent to participate.
* Demonstrate willingness to comply with all study procedures and be available for the study duration.
* Ages 18 to 54 years of age.
* A man.
* Self-report any of the following behaviors and/or health conditions

  1. Diagnosed with bacterial sexually transmitted infection (e.g., syphilis, gonorrhea, or chlamydia)
  2. Sex with a partner who is living with HIV
  3. Sex without a condom with two or more partners whose HIV status were unknown
  4. Injection drug use and sharing injection equipment
* Have been without a PrEP prescription for at least 24 weeks.

Exclusion Criteria:

* Diminished capacity to consent due to:

  1. Inability to provide informed consent (e.g., cognitive impairment), or
  2. Presence of severe psychiatric symptoms (e.g., mania, psychosis) that impair the ability to provide informed consent, as assessed by interviewers trained in CITI Human Subjects Research and NIH Good Clinical Practice.
* Younger than 18 or older than 54 years of age.
* A woman.
* Does not self-report any of the following behaviors and/or health conditions

  1. Diagnosed with bacterial sexually transmitted infection (e.g., syphilis, gonorrhea, or chlamydia)
  2. Sex with a partner who is living with HIV
  3. Sex without a condom with two or more partners whose HIV status were unknown
  4. Injection drug use and sharing injection equipment
* Has had an active PrEP prescription within the past 24 weeks.
* Living with HIV (e.g. has received an HIV diagnosis).
* Planning to move outside of Miami-Dade or Broward counties in the next 7 months.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Self-report attendance at first PrEP appointment | Baseline, 3 months, and 6 months
  Attendance at the first scheduled PrEP (pre-exposure prophylaxis) appointment will be assessed using self-report responses at baseline, 3 months, and 6 months. Participants will respond to the question: "Did you attend your first scheduled PrEP appointment?" with binary options (Yes/No). This will be measured by the percentage of participants responding "Yes" at each time point and will evaluate engagement with PrEP services over time.

SECONDARY OUTCOMES:
PrEP Cascade Questionnaire, measured by participant survey responses | Baseline, 3 months, and 6 months
  The PrEP Cascade Questionnaire is a structured survey designed to assess participant engagement across stages of the PrEP prevention cascade (awareness, access, initiation, adherence, and retention). Each item will be scored as binary (Yes/No) or categorical (e.g., aware/not aware, initiated/not initiated, adherent/non-adherent). This will be measured by the percentage of participants meeting each cascade stage at each time point and will evaluate the progression through the PrEP cascade over time.
Percentage of correct PrEP questions, measured by participant survey responses | Baseline, 3 months, and 6 months.
  The PrEP Questionnaires is a structured survey designed to assess participant PrEP knowledge. Each item will be scored as binary (Yes/No) or categorical. This will be measured by the percentage of correct responses at each time point and will evaluate PrEP knowledge over time.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano R Kanamori, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States